CLINICAL TRIAL: NCT04993560
Title: Comparing the Safety and Efficacy of Homologous and Heterologous COVID-19 Prime-boost Vaccination in Bahrain
Brief Title: Safety and Efficacy of COVID-19 Prime-boost Vaccine in Bahrain
Status: Completed | Type: Observational
Sponsor: Royal College of Surgeons in Ireland - Medical University of Bahrain (Other)
Collaborators: The National Taskforce for Combatting COVID-19- Kingdom of Bahrain (Unknown); Bahrain Defence Force Royal Medical Services (Unknown); Ministry of Health, Bahrain (Other Government); Bahrain International Exhibition & Convention Centre (Unknown)
Responsible Party: Sponsor
Other Study IDs: CRT- COVID2021-143
Record Dates: First submitted 2021-08-04; First posted 2021-08-06 (Actual); Last update posted 2021-10-26 (Actual); Status verified 2021-08

CONDITIONS: SARS-CoV 2 Infection; Covid19
Keywords: Safety; Efficacy; Prime-boost vaccine; COVID-19; BBIBP-CorV booster; BNT162b2 booster
MeSH Terms: conditions — COVID-19 | interventions — BIBP COVID-19 vaccine; BNT162 Vaccine

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Homologous booster: Two doses of BBIBP-CorV, followed by BBIBP-CorV
  Interventions: Biological: BBIBP-CorV
- Heterologous booster: Two doses of BBIBP-CorV, followed by BNT162b2
  Interventions: Biological: BNT162b2

INTERVENTIONS:
Biological: BBIBP-CorV — Inactivated virus COVID-19 vaccine
  Other Names: Sinopharm COVID-19 vaccine
  Groups: Homologous booster
Biological: BNT162b2 — mRNA-based COVID-19 vaccine
  Other Names: Pfizer-BioNTech vaccine
  Groups: Heterologous booster

SUMMARY:
Coronavirus disease 2019 (COVID-19) is potentially a deadly disease caused by severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) that targets the lung mainly, resulting in respiratory tract infections in humans. It has developed into a pandemic with serious global public health problems.

Recent research has shown that the new SARS-CoV-2 variants reduces the efficacy of the vaccinations and are predominantly more transmissible or infective. A few countries namely Bahrain, United Arab Emirates, and Turkey have recently started introducing a booster dose following primary two doses of the COVID-19 immunization series.

This study aims to identify which booster dose is more effective; taking a booster dose from the same vaccine initially taken or a booster dose from a different vaccine than initially taken.

DETAILED DESCRIPTION:
According to the World Health Organization COVID-19 Dashboard, the coronavirus disease 2019 pandemic, has caused over 181 million infections and more than 3 million deaths worldwide as of July 1, 2021. COVID-19 is potentially a deadly disease caused by severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) that targets the lung mainly resulting in respiratory tract infections in humans. This has become a serious concern for public health.

Among the currently approved COVID-19 vaccines in the Kingdom of Bahrain, BBIBP-CorV (inactivated virus) vaccine and BNT162b2 (mRNA vaccine) is being administered to the population.

Inactivated vaccines have been extensively studied. In a phase 1/2 trial, the BBIBP-CorV vaccine has shown to be generally safe against COVID-19 and induce antibody responses. However, WHO's Strategic Advisory Group of Experts (SAGE) experts have summarized information from clinical trials in Bahrain, United Arab Emirates, Egypt, Jordan, and China indicating that individuals with comorbidities and older adults (≥60 years) who received 2 doses of BBIBP-CorV have low confidence in the efficacy of preventing COVID-19.

Current clinical trials have played a key role in the approval of different COVID vaccines based on their efficacy data, however, there is still uncertainty regarding the duration of protection from these vaccines towards the COVID -19 virus. Recent evidence has shown that the new SARS-CoV-2 variants reduces the efficacy of the vaccinations and are predominantly more transmissible or infective.

A few countries namely Bahrain, United Arab Emirates, and Turkey have recently started introducing a booster dose following primary two doses of the COVID-19 immunization series. The enhanced humoral response has been seen in homologous vaccination. Heterologous vaccination has shown to significantly induce more immunogenicity than homologous vector boost, and higher or comparable to the homologous mRNA regimens. Strong humoral and immune response has also been induced by heterologous vector-mRNA boosting with an acceptable reactogenicity profile.

To our knowledge, there has been no research conducted to date on the reactogenic and immunogenetic response of a COVID-19 booster dose after completing the primary two doses of the COVID-19 immunization series. This study will compare the reactogenic and immunogenetic response of heterologous BNT162b2 booster dose after completing two doses of BBIBP-CorV vaccination versus homologous BBIBP-CorV booster after completing two doses of BBIBP-CorV vaccination.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged ≥21yo.
* Asymptomatic 24h before the administration of booster dose.
* Has no active or previous RT-PCR lab-confirmed COVID-19 diagnosis.
* Completed three months to six months after the second dose of BBIBP-CorV.
* Have at least one Antibody test done before receiving the BBIBP-CorV booster dose OR can be done if the participant is yet to receive the BNT162b2 booster dose.
* Tested negative using Rapid Antigen Detection Test on the day of receiving the booster (positive results will confirm with RT-PCR).
* Study participants must have the ability to give informed consent.

Exclusion Criteria:

* Children aged <21yo.
* Symptomatic within 24h before the administration of booster dose.
* Has active or previous RT-PCR lab-confirmed COVID-19 diagnosis.
* Did not complete three months to six months after the second dose of BBIBP-CorV.
* Does not have at least one Antibody test done before receiving the BBIBP-CorV booster dose
* Tested positive using Rapid Antigen Detection Test on the day of receiving the booster (positive results will be confirmed with PCR).
* Patients unable to give informed consent.

Min Age: 21 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Adults aged ≥21yo. Asymptomatic 24h before the administration of booster dose. Has no active or previous RT-PCR lab-confirmed COVID-19 diagnosis. Tested negative using Rapid Antigen Detection Test on the day of receiving the booster
Sampling Method: Probability Sample
Enrollment: 305 (Actual)
Dates: Start 2021-07-18 (Actual); Primary Completion 2021-09-17 (Actual); Study Completion 2021-10-19 (Actual)

PRIMARY OUTCOMES:
Change from Baseline Immunogenicity at 8 weeks | before the reception of the booster dose and on the 8th week after the reception of the booster dose
  Antigen-specific humoral immune response will be analyzed using one commercial immunoassay (S, N) and one pseudovirus neutralization assay (sVNT)

SECONDARY OUTCOMES:
Reactogenicity | A follow-up call will be made to participants that received booster doses on day 1 and day 5. To review any adverse events a weekly phone call will be made for a total of 8 weeks from the date of recruitment.
  The intensity of adverse events will be graded according to a 4-grade scale:
  Grade 1 (mild), Grade 2 (moderate), Grade 3 (severe), and Grade 4 (life-threatening).
  Reactogenicity symptoms can be:
  Local: (Hardness, Itch, Pain, Warmth, Redness, and Swelling)
  • Systemic: (Chills, Fatigue, Fever, Feverish, Headache, Joint pain, Malaise, Muscle ache, Nausea, Vomiting, Diarrhea)

CONTACTS AND LOCATIONS:
Overall Officials: Manaf AlQahtani, Dr., Principal Investigator — Royal College of Surgeons in Ireland - Bahrain
Locations (1):
- Royal College of Surgeons in Ireland - Bahrain, Manama, Bahrain

IPD SHARING:
Plan to Share IPD: Yes
Monitoring, audits, and Research Ethics Committee review will be permitted and provide direct access to source data and documents. The Lead PI and the researchers assigned by him will have access to the stored data/specimens. Only the Lead PI and the researchers assigned working on this study will be eligible to obtain the data/specimens from the participants during data collection.
Supporting Information: Study Protocol, SAP, CSR, Analytic Code
Time Frame: Dr Manaf will act as the data custodian and is responsible for the storage, handling and quality of the study data.
  Data will be collected in the case report form to allow for cross referencing to check validity.
  Study documents (paper and electronic) will be retained in a secure (kept locked when not in use) location during and after the trial has finished. All essential documents including source documents will be retained for a period of 5 years after study completion (last patient, last study point). A label stating the date after which the documents can be destroyed will be placed on the inside front cover of the case notes of trial participants.
Access Criteria: Study documents (paper and electronic) will be retained in a secure (kept locked when not in use) location during and after the trial has finished.

REFERENCES:
- [Background] Chen N, Zhou M, Dong X, Qu J, Gong F, Han Y, Qiu Y, Wang J, Liu Y, Wei Y, Xia J, Yu T, Zhang X, Zhang L. Epidemiological and clinical characteristics of 99 cases of 2019 novel coronavirus pneumonia in Wuhan, China: a descriptive study. Lancet. 2020 Feb 15;395(10223):507-513. doi: 10.1016/S0140-6736(20)30211-7. Epub 2020 Jan 30. PMID 32007143
- [Background] Wang C, Horby PW, Hayden FG, Gao GF. A novel coronavirus outbreak of global health concern. Lancet. 2020 Feb 15;395(10223):470-473. doi: 10.1016/S0140-6736(20)30185-9. Epub 2020 Jan 24. No abstract available. PMID 31986257
- [Background] WHO Coronavirus (COVID-19) Dashboard [Internet]. World Health Organization. World Health Organization; [cited 2021Jul1]. Available from: https://covid19.who.int/
- [Background] Xia S, Zhang Y, Wang Y, Wang H, Yang Y, Gao GF, Tan W, Wu G, Xu M, Lou Z, Huang W, Xu W, Huang B, Wang H, Wang W, Zhang W, Li N, Xie Z, Ding L, You W, Zhao Y, Yang X, Liu Y, Wang Q, Huang L, Yang Y, Xu G, Luo B, Wang W, Liu P, Guo W, Yang X. Safety and immunogenicity of an inactivated SARS-CoV-2 vaccine, BBIBP-CorV: a randomised, double-blind, placebo-controlled, phase 1/2 trial. Lancet Infect Dis. 2021 Jan;21(1):39-51. doi: 10.1016/S1473-3099(20)30831-8. Epub 2020 Oct 15. PMID 33069281
- [Background] https://cdn.who.int/media/docs/default-source/immunization/sage/2021/april/2_sage29apr2021_critical-evidence_sinopharm.pdf
- [Background] Moore JP, Offit PA. SARS-CoV-2 Vaccines and the Growing Threat of Viral Variants. JAMA. 2021 Mar 2;325(9):821-822. doi: 10.1001/jama.2021.1114. No abstract available. PMID 33507218
- [Background] Li Q, Wu J, Nie J, Zhang L, Hao H, Liu S, Zhao C, Zhang Q, Liu H, Nie L, Qin H, Wang M, Lu Q, Li X, Sun Q, Liu J, Zhang L, Li X, Huang W, Wang Y. The Impact of Mutations in SARS-CoV-2 Spike on Viral Infectivity and Antigenicity. Cell. 2020 Sep 3;182(5):1284-1294.e9. doi: 10.1016/j.cell.2020.07.012. Epub 2020 Jul 17. PMID 32730807
- [Background] Li Q, Nie J, Wu J, Zhang L, Ding R, Wang H, Zhang Y, Li T, Liu S, Zhang M, Zhao C, Liu H, Nie L, Qin H, Wang M, Lu Q, Li X, Liu J, Liang H, Shi Y, Shen Y, Xie L, Zhang L, Qu X, Xu W, Huang W, Wang Y. SARS-CoV-2 501Y.V2 variants lack higher infectivity but do have immune escape. Cell. 2021 Apr 29;184(9):2362-2371.e9. doi: 10.1016/j.cell.2021.02.042. Epub 2021 Feb 23. PMID 33735608
- [Background] Ramshaw IA, Ramsay AJ. The prime-boost strategy: exciting prospects for improved vaccination. Immunol Today. 2000 Apr;21(4):163-5. doi: 10.1016/s0167-5699(00)01612-1. No abstract available. PMID 10740236
- [Background] Shaw RH, Stuart A, Greenland M, Liu X, Nguyen Van-Tam JS, Snape MD; Com-COV Study Group. Heterologous prime-boost COVID-19 vaccination: initial reactogenicity data. Lancet. 2021 May 29;397(10289):2043-2046. doi: 10.1016/S0140-6736(21)01115-6. Epub 2021 May 12. No abstract available. PMID 33991480
- [Background] Schmidt T, Klemis V, Schub D, Mihm J, Hielscher F, Marx S, et al. Immunogenicity and reactogenicity of a heterologous COVID-19 prime-boost vaccination compared with homologous vaccine regimens. 2021;
- [Background] Gross R, Zanoni M, Seidel A, Conzelmann C, Gilg A, Krnavek D, Erdemci-Evin S, Mayer B, Hoffmann M, Pohlmann S, Liu W, Hahn BH, Beil A, Kroschel J, Jahrsdorfer B, Schrezenmeier H, Kirchhoff F, Munch J, Muller JA. Heterologous ChAdOx1 nCoV-19 and BNT162b2 prime-boost vaccination elicits potent neutralizing antibody responses and T cell reactivity against prevalent SARS-CoV-2 variants. EBioMedicine. 2022 Jan;75:103761. doi: 10.1016/j.ebiom.2021.103761. Epub 2021 Dec 17. PMID 34929493
- [Derived] Mallah SI, Alawadhi A, Jawad J, Wasif P, Alsaffar B, Alalawi E, Mohamed AM, Butler AE, Alalawi B, Qayed D, Almahari SA, Mubarak A, Mubarak A, Saeed S, Humaidan A, Kumar N, Atkin S, Alqahtani M. Safety and efficacy of COVID-19 prime-boost vaccinations: Homologous BBIBP-CorV versus heterologous BNT162b2 boosters in BBIBP-CorV-primed individuals. Vaccine. 2023 Mar 17;41(12):1925-1933. doi: 10.1016/j.vaccine.2023.01.032. Epub 2023 Jan 23. PMID 36725431